CLINICAL TRIAL: NCT05784662
Title: Evaluating the Social Workers Addressing Firearm Risk (SAFR) Intervention: A Pilot Study
Brief Title: Social Workers Addressing Firearm Risk
Acronym: SAFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Patricia Logan-Greene, Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00006636; UL1TR001412 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-03-27 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Gun Violence Prevention
Keywords: firearms; guns; social work

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Workers Addressing Firearm Risk (Experimental): The Social workers Addressing Firearm Risk (SAFR) intervention is fully-online intervention that contains four modules. Each module includes interviews with experts, didactic content, handouts, and brief quizzes to check learning (required by New York State for continuing education credit).
  Interventions: Behavioral: Social Workers Addressing Firearm Risk
- Control (No Intervention): Wait list control. Will receive access to SAFR intervention at conclusion of the study.

INTERVENTIONS:
Behavioral: Social Workers Addressing Firearm Risk — Educational intervention for social workers.
  Other Names: SAFR
  Arms: Social Workers Addressing Firearm Risk

SUMMARY:
Aim 2: Evaluate the preliminary efficacy of the SAFR intervention using a randomized controlled trial. An additional 100 practicing social workers (excluding participants from Aim 1) will be recruited, with n = 50 allocated to each arm of the study utilizing block randomization. Participants in the control arm will receive invitations to all surveys but not to the SAFR intervention itself. We will utilize the validated measures from Aim 1 to assess changes on study variables. Results will be analyzed using either mixed linear models or generalized estimating equations as appropriate. Analyses will be performed with a focus on estimation of parameters for use in the planning of a subsequent comparative trial designed to fully assess intervention efficacy with a national sample. Supportive analyses that adjust for participant covariates will also be considered. We will also ask participants for feedback on the intervention and will track indicators of feasibility and acceptability (recruitment rates, completion of intervention and measurement tools).

DETAILED DESCRIPTION:
Specific Aim 2: Evaluate the efficacy of the SAFR intervention. Once measurement tools have been validated, we will begin to recruit for the pilot test of the SAFR intervention. Recruitment methods will be similar to those in Aim 1; individuals who participate in Aim 1 will not be eligible to participate in the trial of SAFR. Participants will be randomized equally to the control and intervention groups. Participants will be invited to enroll in the study by clicking on links in advertisement materials. The link will take them to a brief webpage with information about the study and questions screening for eligibility. Once screened, they will complete the informed consent document and await randomization. Participants in the intervention group will receive an email with instructions on how to access the pre-test measurements and the course. Because the course is online and self-paced, they will be given six weeks to complete the course, with reminders coming once a week to encourage completion. The UB SSW Continuing Education website allows us to track information about participants, including time to completion for all users; this information will be utilized to assess the acceptability of the course. The pre-test survey will include the scales assessing knowledge, attitudes, and behaviors towards assessing for risks of firearm violence among clients, in addition to a demographic survey and the Gun Control Attitudes and Gun Behaviors and Beliefs Scales. The post-test, which will be sent out one month after the pre-test, assuming that the course was successfully completed, will contain the measures regarding knowledge, attitudes, and behaviors. We will also be assessing for acceptability of the intervention by including questions that ask participants for their thoughts on the course. Finally, the follow-up will be sent three months after the completion of the post-test and will assess knowledge, attitudes, and behaviors a final time. The control group will receive the three surveys (without course feedback items) on the same timeline. At the conclusion of the study, they will be invited to receive the SAFR intervention at no cost.

Data analysis plan. To describe the observed variability in the data and test for differences between randomized groups, linear or generalized linear models will be utilized depending on the nature of the outcome. Once a given model is fit, a linear contrast based on the estimated model parameters will be constructed and used to test for the overall effect of random assignment. Point estimates and corresponding confidence intervals to quantify treatment differences will be provided. Since the comparability of randomized groups may be questioned due to chance imbalances in confounding variables, subject-level covariates known to be predictive of outcome and their interactions with randomized assignment will be added to the models as a series of supportive analyses. All analyses will be performed based on the intent-to-treat principle. The amount and nature of missing data for collected study variables will be characterized and no method of imputation will be used for missing data for primary analyses. All tests will be two-sided and tested at a 0.05 nominal significance level. Standard diagnostic plots will be used to assess model fit and transformations of variables may be considered in order to meet statistical assumptions. With the proposed sample size, mean differences of 0.6 standard deviations are detectable at 80% power. Group-specific means and proportions will be estimated with an associated confidence interval width of 0.55 standard deviations and 28 percentage points, respectively.

Hypotheses:

Aim 2: The SAFR intervention will improve social workers' knowledge of gun violence, attitudes about social workers' need to intervene with all clients, and behaviors regarding discussing guns and gun violence risks with clients compared to pre-test and the control group. We also hypothesize that the SAFR intervention will be feasible and acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Practicing social worker
* In New York
* Age 18 or older
* English proficiency

Exclusion Criteria:

* Not meeting above criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Online Only, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- SAFR Arm: Proportion of the randomized sample that received the SAFR intervention, a self-paced 4 hour online training about how to assess and intervene with clients at-risk for gun violence.
- WL Control Arm: Proportion of the randomized sample that did not receive the SAFR intervention during the study period.
Period: Overall Study
Arm/Group | SAFR Arm | WL Control Arm
Started | 63 | 48
Completed | 42 | 31
Not Completed | 21 | 17
Not completed — Lost to Follow-up | 21 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Workers Addressing Firearm Risk | Control | Total
Number analyzed (Participants) | 63 | 48 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 47 | 107
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (10.9) | 39.7 (11.2) | 40.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 46 | 34 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 52 | 41 | 93
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 48 | 111

OUTCOME MEASURES:

1. Primary Outcome: Change in Knowledge About Gun Violence
Description: Assessed with the Knowledge about gun violence measure (novel). Theoretical minimum/maximum = 0.0/5.0. High scores indicate more knowledge about firearm safety.
Time Frame: Baseline, 1 month later, and 3 months later
Population: Some participants lost to follow up and/or had missing data on outcomes measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SAFR Arm: Proportion of the randomized sample that received the SAFR intervention.
Arm/Group | SAFR Arm | WL Control Arm
Number analyzed (Participants) | 47 | 38
score on a scale
  Baseline (pretest) | 2.49 (0.47) | 2.54 (0.56)
  One month later (post-test): number analyzed (Participants) | 46 | 38
  One month later (post-test) | 2.94 (0.48) | 2.66 (0.48)
  Three months later (follow-up): number analyzed (Participants) | 42 | 32
  Three months later (follow-up) | 3.01 (0.45) | 2.63 (0.59)

2. Primary Outcome: Change in Attitudes About Firearms Safety Counseling
Description: Assessed with the Attitudes about firearms safety counseling (novel). Theoretical minimum/maximum = 0/5.00. High scores indicate greater inclination towards discussing firearm safety with clients.
Time Frame: Baseline, 1 month later, and 3 months later
Population: Some participants lost to follow up and/or had missing data in outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAFR Arm | WL Control Arm
Number analyzed (Participants) | 63 | 48
score on a scale
  Baseline (pre-test) | 2.97 (0.50) | 3.09 (0.44)
  One month later (post-test): number analyzed (Participants) | 46 | 38
  One month later (post-test) | 3.14 (0.48) | 3.13 (0.44)
  Three months later (follow-up): number analyzed (Participants) | 42 | 31
  Three months later (follow-up) | 3.25 (0.43) | 3.11 (0.52)

3. Primary Outcome: Change in Confidence About Firearms Safety Counseling
Description: Assessed with the Confidence about firearms safety counseling (novel). Theoretical minimum/maximum = 0/5.00. High scores indicate greater confidence about discussing firearm safety with clients.
Time Frame: Baseline, 1 month later, and 3 months later
Population: Some participants lost to follow up and/or had missing data on outcomes measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SAFR Arm | WL Control Arm
Number analyzed (Participants) | 52 | 40
units on a scale
  Baseline (pre-test) | 2.41 (0.75) | 2.41 (0.84)
  One month later (post-test): number analyzed (Participants) | 46 | 38
  One month later (post-test) | 2.91 (0.73) | 2.65 (0.66)
  Three months later (follow-up): number analyzed (Participants) | 41 | 31
  Three months later (follow-up) | 3.01 (0.66) | 2.70 (0.76)

4. Primary Outcome: Change in Behaviors With Clients
Description: Assessed with the Behaviors with Clients measure (novel). Theoretical minimum/maximum = 0/5.00. High scores indicate more interventions about firearm safety with clients. This scale asked questions like, "I talk to my clients about firearm access," with answers ranging from Strongly disagree to strongly agree.
Time Frame: Baseline, 1 month later, and 3 months later
Population: Some participants lost to follow up and/or had missing data on outcomes measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SAFR Arm | WL Control Arm
Number analyzed (Participants) | 52 | 39
units on a scale
  Baseline (pre-test) | 2.07 (0.74) | 2.13 (0.82)
  One month later (post-test): number analyzed (Participants) | 45 | 37
  One month later (post-test) | 2.44 (0.44) | 2.23 (0.76)
  Three months later (follow-up): number analyzed (Participants) | 39 | 30
  Three months later (follow-up) | 2.64 (0.66) | 2.31 (0.74)

5. Primary Outcome: Change in Behaviors With Clients in Last Month
Description: Assessed with the Behaviors with Clients in last month measure (novel). Theoretical minimum/maximum = 0/2.00. Higher scores indicate more interventions about firearm safety with clients. This scale asked questions like, "In the last month, I have provided clients with information about firearm safety..." with answers specified as "none of the time," "some of the time," and "all of the time."
Time Frame: Baseline, 1 month later, and 3 months later
Population: Some participants lost to follow up and/or had missing data on outcomes measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SAFR Arm | WL Control Arm
Number analyzed (Participants) | 53 | 43
units on a scale
  Baseline (pre-test) | 0.77 (0.52) | 0.74 (0.51)
  One month later (post-test): number analyzed (Participants) | 46 | 38
  One month later (post-test) | 0.91 (0.56) | 0.86 (0.51)
  Three months later (follow-up): number analyzed (Participants) | 42 | 29
  Three months later (follow-up) | 0.93 (0.59) | 0.97 (0.53)

ADVERSE EVENTS:
Time Frame: Approximately 9 months
Description: Definitions did not differ. All research team members watched for signs of adverse events during the study timeline. Additionally, participants were provided with contact information for the study team in case an adverse event occured.
Arm/Group | SAFR Arm | WL Control Arm
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/48
Other Adverse Events (participants affected / at risk) | 0/63 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT05784662/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT05784662/ICF_001.pdf